CLINICAL TRIAL: NCT01428206
Title: Liverpool Care Pathway for the Dying at Residential Care Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Margareta Brännström, RNT/PHD, Umeå University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCP001
Record Dates: First submitted 2011-08-23; First posted 2011-09-02 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: End-of-life Care
Keywords: palliative care; nursing homes; Liverpool care pathway
MeSH Terms: interventions — Terminal Care; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liverpool care pathway (Other): Liverpool care pathway for dying at nursing homes
  Interventions: Other: Liverpool care pathway
- control (No Intervention): Usual care is performed for the control group

INTERVENTIONS:
Other: Liverpool care pathway — Liverpool care pathway is started tha last day in life for elderly at nursing homes
  Other Names: end-of-life care; palliative care
  Arms: Liverpool care pathway

SUMMARY:
Liverpool Care Pathway for the dying patient (LCP) was developed to transfer the care practice from the hospice setting to the hospital setting in UK. LCP is a pathway with standardized registration method to monitor the care and its results. The primary aim is to study the effects of LCP on dying patients symptom burden and communication with close relatives and health care professionals.

DETAILED DESCRIPTION:
All residential care homes in Skellefteå municipality are included in the study and randomized either to control or intervention group. During the baseline period the care is provided as usual. During the intervention period the LCP is used for patients for whom the dying phase is diagnosed in the intervention group. Usual care is performed for the control group. After death of a patient a close relative fill in a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* nursing homes in Skellefteå municipality, Sweden

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
quality of care | one month to six months after the relatives death
  changes between the groups about values of symptom scores on the Edmonton assessment scale (ESAS) and the views of informal carers-evaluation of services (VOICES)assessed by close relative

SECONDARY OUTCOMES:
place of death | the time of death
  changes between the groups
drug consumption | the last three days before death

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Brännström, PhD, Principal Investigator — Department of nursing, Umeå University
Locations (1):
- Skellefteå municipality, Skellefteå, Västerbotten County, Sweden